CLINICAL TRIAL: NCT02695979
Title: Changes of Macrophage Migration Inhibitory Factor and Thyroid Hormones During Liver Transplantation. Association With Graft Dysfunction
Brief Title: Changes of Macrophage Migration Inhibitory Factor During Orthotopic Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Joanna Stefaniak, Dr.med., Medical University of Vienna
Other Study IDs: 1458/2014
Record Dates: First submitted 2016-01-12; First posted 2016-03-02 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Evidence of Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, graft liver effluent, urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing OLT: Patients aged 18-70 with end-stage liver disease undergoing orthotopic liver transplantation (OLT).

SUMMARY:
Collecting blood, graft liver effluent and urine samples from patients undergoing orthotopic liver transplantation.

DETAILED DESCRIPTION:
Aims are to measure Macrophage Migration Inhibitory Factor, Macrophage Migration Inhibitory Factor II and its' soluble receptor CD74 in serum, liver graft effluent and urine in and evaluate MIF's role in hepatic ischemia/reperfusion injury, postoperative graft function and kidney function.

ELIGIBILITY:
Inclusion Criteria:

* End stage liver disease, chronic liver failure, orthotopic liver transplantation

Exclusion Criteria:

* Combined transplantations (liver plus kidney or lung), age under 18 y, acute liver failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing orthotopic liver transplantation
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2018-09 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Macrophage Migration Inhibitory Factor in human serum, liver graft effluent and urine | 24 months

OTHER OUTCOMES:
Acute kidney injury, outcome | 48 months
  Acute kidney injury, outcome

CONTACTS AND LOCATIONS:
Overall Officials: Peter Faybik, Prof, Study Chair — Medical University Vienna, Department of Anesthesia, General Intensive Care and Pain Management
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No